CLINICAL TRIAL: NCT03159234
Title: Evaluation of New Methods for Prediction of Fetal Lung Maturity in Diabetic Mothers
Brief Title: Prediction of Fetal Lung Maturity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer of obstetrics and gynecology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17100188
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Fetal Distress
MeSH Terms: conditions — Fetal Distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetic pregnant women (Other)
  Interventions: Radiation: fetal lung volume; Radiation: pulmonary artery resistance index; Radiation: Fetal adrenal gland volume:

INTERVENTIONS:
Radiation: fetal lung volume — the best method for measurement of fetal lung volume is by the rotational technique in which each lung is obtained by serial contouring of the pulmonary area after rotating the volumetric image.this is more recent method seems to have advantages allowing finer contouring of the lung and subsequent modification of the contour as well as being better able to estimate the volumes of irregular and small lung as in congenital diaphragmatic hernia
Radiation: pulmonary artery resistance index — Women placed in semirecumbent position and an axial plane through the fetal thorax to achieve 4 chamber view of the heart. The main pulmonary artery was followed to the point where it divides into right and left branches by rotating the transducer from the 4 chamber view to the short axis view of the heart. Pulsed and colour Doppler was used. The fetal pulmonary artery flow waveform measurements was taken within the proximal portion of the main pulmonary artery
Radiation: Fetal adrenal gland volume: — the adrenal gland has a characteristic sonographic appearance; each limb is seen as a long anechoic structure with a thin, echogenic line within its center . Both limbs can sometimes be seen in the coronal plane, and if so there is a strong echogenic line between limbs (probably fat). On the basis of pathologic and histologic studies , we believe the anechoic bulk of the gland represents the fetal zone of the cortex, while the central echogenic core is the medulla.

SUMMARY:
Diabetes is the most common medical complication of pregnancy in the united states four to five percent of pregnancies are complicated by diabetes.

Pregestational diabetes (diabetes diagnosed before pregnancy, type 1 or type 2 diabetes mellitus) comprises approximately 13 percent of all diabetes in pregnancy, while gestational diabetes ( diabetes with onset or first recognition in pregnancy) comprises the remaining 87 percent . The prevalence of pregestational diabetes has been increasing due to the increasing prevalence of type 2 diabetes in women of reproductive age . The mainstay of the medical management of pregestational diabetes involves frequent monitoring of blood glucose levels with adjustment of diet and insulin therapy to achieve normoglycemia. Normoglycemia is important because maintenance of maternal blood glucose concentration at or near normoglycemic levels decreases the likelihood of adverse pregnancy outcomes, such as miscarriage , congenital anomalies , macrosomia and fetal death.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant diabetic women
* 37 weeks gestational age .

Exclusion Criteria:

* Women before 37 and after 39 weeks gestational age
* Pregnancies with known fetal anomalies that may potentially affect the lung maturity .
* Multiple pregnancies.
* Women received steroids for lung maturation after ultrasound image acquisition and before delivery .
* Women with premature rupture of membranes (prom)
* Pregnancies complicated by medical disorders other than diabetes mellitus .
* Failure to obtain an informed consent .

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
APGAR score | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided